CLINICAL TRIAL: NCT00065663
Title: Growth Factor Gene Therapy for Wound Healing
Brief Title: Gene Therapy to Improve Wound Healing in Patients With Diabetes
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Tissue Repair Company (Industry)
Allocation: Non-Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: NIAMS-093; R44AR046154 (NIH)
Record Dates: First submitted 2003-07-30; First posted 2003-07-31 (Estimated); Last update posted 2007-11-20 (Estimated); Status verified 2007-11

CONDITIONS: Wounds and Injuries; Diabetes; Diabetic Foot Ulcers; Foot Wounds
Keywords: gene transfer; adenovirus; platelet-derived growth factor-B; collagen; diabetic ulcer; foot; wounds; diabetic; ulcers
MeSH Terms: conditions — Wounds and Injuries; Diabetes Mellitus; Diabetic Foot; Adenoviridae Infections; Ulcer

INTERVENTIONS:
Genetic: GAM501

SUMMARY:
Patients with diabetes may develop chronic wounds that respond poorly to treatment. Gene therapy with the platelet-derived growth factor-B gene has been shown to help with the healing of chronic wounds. This study will evaluate a new way to deliver the gene to the wound tissue.

DETAILED DESCRIPTION:
Chronic wounds, such as diabetic ulcers, pressure ulcers, and venous stasis ulcers, cause significant morbidity in millions of patients each year in the United States. Individuals with long-standing diabetes develop both peripheral vascular disease and peripheral neuropathy. These patients may not feel pressure from shoes or objects which can damage their skin. Once a wound is formed, it may heal very slowly or not at all due to diabetic complications.

Platelet-derived growth factor-B (PDGF-B) has been approved for use in diabetic ulcers. However, delivery and maintenance of the drug at the wound site in sufficient quantities for a sufficient period of time is a major hurdle to widespread use.

Gene activated matrix (GAM) technology offers the opportunity to place a therapeutic gene contained within a structural matrix into a wound site. This study will evaluate the safety and potential clinical utility of topical applications of GAM501, a gene for PDGF-B contained within an E1-deleted adenoviral vector and formulated in a bovine type I collagen gel. This formulation allows for the migration of wound repair cells into the structural matrix, where they encounter the viral vector and subsequently produce the therapeutic protein within the local wound environment.

Participants in this study will receive up to four treatments with GAM501. Participants will be followed by multiple observations over a 6 to 7 month period.

ELIGIBILITY:
Inclusion Criteria

* Adequately controlled diabetes mellitus (type I or II) as defined by HbA1c < 10.0%
* Cutaneous, lower extremity, plantar medial or lateral surface ulcer between 1 and 10 cm2 post-debridement
* Ulcer present for > 6 weeks prior to study entry
* Ulcer free of all necrotic and infected soft tissue
* Affected limb transcutaneous oxygen pressure (TcpO2) > 30 mmHg at screening or a palpable dorsal pedal or posterior tibial pulse
* Inability to perceive 10 grams pressure using a Semmes-Weinstein 5.07 monofilament in the peri-ulcer area

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21
Dates: Start 2002-08; Study Completion 2004-12

CONTACTS AND LOCATIONS:
Overall Officials: Barbara Sosnowski, PhD, Study Director — Tissue Repair Company
Locations (2):
- United States (2):
  - Foot and Ankle Medical Center, Phoenix, Arizona
  - University of California, San Diego, San Diego, California